CLINICAL TRIAL: NCT01348893
Title: Evaluation of Yoga During School as a Behavioral Prevention Program for Adolescent Health
Brief Title: Evaluation of a Yoga Program in Schools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Kripalu Center for Yoga and Health (Other)
Responsible Party: Principal Investigator, Sat Bir Khalsa, PhD, Assistant Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2007P002600A
Record Dates: First submitted 2010-04-29; First posted 2011-05-06 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Adolescent Development
Keywords: Mental health; Education; Mind Body Therapies
MeSH Terms: conditions — Psychological Well-Being | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical education as usual (No Intervention): High school physical education curriculum established by the school, including competitive sports, aerobic and anaerobic activities, balance and coordination skills. Yoga is not a component of the curriculum.
- Yoga during physical education (Experimental)
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Behavioral: Yoga — 12 to 16 weeks of group yoga classes (approximately 32 classes per student), 30-45 minutes per class, 2-3 times per week, during physical education class. Yoga program includes physical postures and movement, breathing exercises, partner/group games, deep relaxation and meditative techniques.
  Other Names: Kripalu Yoga In The Schools
  Arms: Yoga during physical education

SUMMARY:
The purpose of this preliminary study is to evaluate the effects of a yoga-based program on high school students' psychological health. Results will be used to generate specific hypotheses of how yoga may improve adolescent mental health.

DETAILED DESCRIPTION:
Specific Aims:

1. To evaluate the hypothesis that 12 weeks of yoga during physical education will be acceptable by and feasible with high school students. To test Specific Aim 1, outcomes assessed at both Monument Mountain Regional High School and Waltham High School include: feasibility and acceptance.
2. To evaluate the hypothesis that yoga will improve self-and parent-reported psychosocial well-being including affect, mood, stress and anxiety in high school students, relative to control students taking regular physical education. To test Specific Aim 2, both primary outcomes (affect and mood) will be assessed at both schools. Additional psychosocial well-being outcomes assessed at Monument Mountain Regional High School include: life purpose/satisfaction and self-confidence during stress; self-esteem; parent-reported psychological difficulties; perceived stress; and sleep quality. Additional psychosocial well-being outcomes assessed at Waltham High School include: self-esteem; parent-reported psychological difficulties; and sleep quality.
3. To evaluate the hypothesis that yoga will improve self- and parent-reported self-regulatory skills including resilience, mindfulness, emotion regulation, anger expression, self-esteem and self-confidence relative to physical education controls. Self-regulation outcomes assessed at Monument Mountain Regional High School include: resilience; mindfulness; emotion regulation; control of anger expression; bullying; health behaviors; substance use risk factors; and attention. Self-regulation outcomes assessed at Waltham High School include: resilience; mindfulness; emotion regulation; control of anger expression; substance use risk factors; and attention.

ELIGIBILITY:
Inclusion Criteria:

* Registered for physical education class

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1693 (Actual)
Dates: Start 2008-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in self-reported negative affect and positive affect measured by the 30-item Positive and Negative Affect Schedule for Children (PANAS-C) | Baseline; during intervention after 4 weeks, 8 weeks and 12 weeks; 1 week post-intervention
Change in self-reported mood as measured by: the 30-item Profile of Mood States Short Form (POMS-SF, total and 6 sub-scales), or the 24-item Brunel University Mood Scale (BRUMS, total and 6 sub-scales) | Baseline; 1 week post-intervention

SECONDARY OUTCOMES:
Change in self-reported resilience (ability to adapt) as measured by the 25-item Resilience Scale (RS) | Baseline, 1 week post-intervention
Change in self-reported life purpose/satisfaction and self-confidence during stress, as measured by the 32-item Inventory of Positive Psychological Attitudes (IPPA) | Baseline, 1 week post-intervention
Change in self-reported mindfulness as measured by the 25-item Child Acceptance and Mindfulness Measure (CAMM) | Baseline, 1 week post-intervention
Change in self-reported emotion regulation as measured by the 10-item Emotion Regulation Questionnaire (ERQ, 2 subscales), or the 36-item Difficulties in Emotion Regulation (DERS, 6 sub-scales) | Baseline; during intervention after 4 weeks, 8 weeks and 12 weeks; 1 week post-intervention
Change in self-reported anger expression and control as measured by part 3 of the 35-item State-Trait Anger Expression Inventory (STAXI2-C/A) | Baseline, 1 week post-intervention
Change in self-reported self-esteem as measured by the 10-item Rosenberg Self-Esteem Scale (RSES) | Baseline, 1 week post-intervention
Feasibility and acceptance of the yoga program as measured by: student and parent forms of the 8-item Yoga Evaluation Questionnaire (YEQ), and 30-minute one-on-one qualitative interviews with students | 1 week post-intervention
Change in parent-reported psychological difficulties (total plus 5 sub-scales) as measured by the 25-item Strength and Difficulties Questionnaire (SDQ), parent/teacher form | Baseline, 1 week post-intervention
Change in self-reported stress levels as measured by the 10-item Perceived Stress Scale (PSS) | Baseline, 1 week post-intervention
Change in self-reported sleep as measured by the 19-item Pittsburgh Sleep Quality Index (PSQI) or the 3-item Adolescent Sleep Quality (ASQ) scale | Baseline, 1 week post-intervention
Change in self-reported bullying and victimization by bullying as measured by the 12-item Peer Relations Questionnaire (PRQ) | Baseline, 1 week post-intervention
Change in self-reported physical activity and eating habits as measured by the 8-item Health Behaviors Survey (HBS) | Baseline, 1 week post-intervention
Change in self-reported substance use risk factors as measured by the 45-item UPPS Impulsive Behavior Scale (UPPS), or the 10-item Brief Sensation Seeking Scale with Slater's Addition (BSSS+S2) | Baseline, 1 week post-intervention
Change in attention as measured by: self-report using the 9-item inattention sub-scale of the ADHD Self-Report Scale (ASRS), and a 20-minute O-SPAN task for working memory capacity | Baseline; during intervention after 4 weeks, 8 weeks and 12 weeks; 1 week post-intervention
Change in self-reported stress levels as measured by the 7-Item subscale of the Depression Anxiety Stress Scale (DASS) | Baseline, 1 week post-intervention
Change in self-reported sensation seeking tendencies as measured by the 12 item Brief Sensation Seeking Scale and Slater's Addition (BSSS+SS2). | Baseline, 1 week post-intervention
Change in self-reported sadness levels as measured by the 3-Item subscale of the Sadness Management Scale (SMS) | Baseline, 1 week post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sat Bir S Khalsa, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (3):
- United States (3):
  - Boston Latin Public School, Boston, Massachusetts
  - Monument Mountain Regional High School, Great Barrington, Massachusetts
  - Waltham Senior High School, Waltham, Massachusetts

REFERENCES:
- [Result] Noggle JJ, Steiner NJ, Minami T, Khalsa SB. Benefits of yoga for psychosocial well-being in a US high school curriculum: a preliminary randomized controlled trial. J Dev Behav Pediatr. 2012 Apr;33(3):193-201. doi: 10.1097/DBP.0b013e31824afdc4. PMID 22343481
- [Result] Khalsa SR, McCarthy KS, Sharpless BA, Barrett MS, Barber JP. Beliefs about the causes of depression and treatment preferences. J Clin Psychol. 2011 Jun;67(6):539-49. doi: 10.1002/jclp.20785. Epub 2011 Mar 1. PMID 21365652
- [Derived] Conboy LA, Noggle JJ, Frey JL, Kudesia RS, Khalsa SB. Qualitative evaluation of a high school yoga program: feasibility and perceived benefits. Explore (NY). 2013 May-Jun;9(3):171-80. doi: 10.1016/j.explore.2013.02.001. PMID 23643372